CLINICAL TRIAL: NCT02620813
Title: De Novo Lipogenesis of Sebaceous Glands in Acne
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 725019
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Acne Vulgaris
Keywords: acne; sebaceous gland; lipid; sebum
MeSH Terms: conditions — Acne Vulgaris | interventions — Tretinoin; Isotretinoin

ARMS (3):
- No Acne (No Intervention): Healthy subjects without acne between the ages of 15-45
- Acne Subjects on Topical Tretinoin Treatment (Experimental): Subjects with acne before and after topical retinoid therapy
  Interventions: Drug: Tretinoin
- Acne Subjects on Systemic Isotretinoin Treatment (Experimental): Subjects with acne before and after isotretinoin therapy
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: Tretinoin — Subjects will apply 0.5% tretinoin cream nightly to their face for a total of 12 weeks.
  Other Names: Retin-A
  Arms: Acne Subjects on Topical Tretinoin Treatment
Drug: Isotretinoin — Subjects will take isotretinoin as prescribed by their dermatologist.
  Arms: Acne Subjects on Systemic Isotretinoin Treatment

SUMMARY:
There are two purposes of this study:

1. First, the investigators want to see what the differences are in de novo sebaceous lipid production of people with and without acne.
2. Secondly, the investigators want to know what happens to sebaceous gland de novo lipid production before and after treatment with topical tretinoin and oral isotretinoin.

DETAILED DESCRIPTION:
The primary objective of this study is to understand how de novo lipid production of sebaceous glands are altered in acne and with acne directed therapy.

Hypothesis 1: The overall de novo lipogenesis will be increased in those with acne

Hypothesis 2: Treatment with topical tretinoin and systemic isotretinoin will reduce de novo lipogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 to 45 years of age
* Subject/Parents/Legal Guardian be able to read and comprehend study procedure and consent forms
* Have acne that is diagnosed by a board certified dermatologist
* Meet one of the following criteria:

  * already been prescribed oral isotretinoin for treatment of acne
  * have already been prescribed a topical retinoid
  * eligible for prescription of topical tretinoin

Exclusion Criteria:

* Those who have already initiated or completed a course of systemic isotretinoin
* Those with seborrheic dermatitis, rosacea, or polycystic ovary syndrome
* Those who are pregnant in female participants
* Those who do not fit the inclusion criteria

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10-12 (Actual); Study Completion 2017-10-12 (Actual)

PRIMARY OUTCOMES:
Sebumeter measurement differences before and after treatment with isotretinoin | 3 months
Change in the fractional contribution of DNL to the total sebum palmitate before and after treatment with isotretinoin at baseline and 3 months after treatment. | 3 months

SECONDARY OUTCOMES:
Change in the global acne grade score | 3 months
Change in the investigator global assessment of acne | 3 months
Change in the lesion counts of inflammatory and non-inflammatory lesions. | 3 months
Difference in the fractional contribution of de novo lipogenesis (DNL) to the sebum total palmitate between those with and without acne | 3 months
Difference in the fractional contribution of DNL to the sebum total palmitate before and after treatment with a topical retinoid (adapalene, tazarotene, or tretinoin). | 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dermatology Research Area, Davis, California
  - UC Davis Department of Dermatology, Sacramento, California

REFERENCES:
- [Background] Rush EC, Chhichhia P, Kilding AE, Plank LD. Water turnover in children and young adults. Eur J Appl Physiol. 2010 Dec;110(6):1209-14. doi: 10.1007/s00421-010-1621-5. Epub 2010 Aug 24. PMID 20734057
- [Background] Blume U, Verschoore M, Poncet M, Czernielewski J, Orfanos CE, Schaefer H. The vellus hair follicle in acne: hair growth and sebum excretion. Br J Dermatol. 1993 Jul;129(1):23-7. doi: 10.1111/j.1365-2133.1993.tb03306.x. PMID 8369207
- [Background] Zouboulis CC, Baron JM, Bohm M, Kippenberger S, Kurzen H, Reichrath J, Thielitz A. Frontiers in sebaceous gland biology and pathology. Exp Dermatol. 2008 Jun;17(6):542-51. doi: 10.1111/j.1600-0625.2008.00725.x. PMID 18474083
- [Background] Thody AJ, Shuster S. Control and function of sebaceous glands. Physiol Rev. 1989 Apr;69(2):383-416. doi: 10.1152/physrev.1989.69.2.383. PMID 2648418
- [Background] Pappas A, Johnsen S, Liu JC, Eisinger M. Sebum analysis of individuals with and without acne. Dermatoendocrinol. 2009 May;1(3):157-61. doi: 10.4161/derm.1.3.8473. PMID 20436883
- [Background] Nakase K, Nakaminami H, Takenaka Y, Hayashi N, Kawashima M, Noguchi N. Relationship between the severity of acne vulgaris and antimicrobial resistance of bacteria isolated from acne lesions in a hospital in Japan. J Med Microbiol. 2014 May;63(Pt 5):721-728. doi: 10.1099/jmm.0.067611-0. Epub 2014 Feb 12. PMID 24523159
- [Background] Thiboutot D, Dreno B, Gollnick H, Bettoli V, Kang S, Leyden JJ, Shalita A, Torres V; Global Alliance to Improve Outcomes in Acne. A call to limit antibiotic use in acne. J Drugs Dermatol. 2013 Dec;12(12):1331-2. No abstract available. PMID 24301232
- [Background] Iinuma K, Sato T, Akimoto N, Noguchi N, Sasatsu M, Nishijima S, Kurokawa I, Ito A. Involvement of Propionibacterium acnes in the augmentation of lipogenesis in hamster sebaceous glands in vivo and in vitro. J Invest Dermatol. 2009 Sep;129(9):2113-9. doi: 10.1038/jid.2009.46. Epub 2009 Mar 12. PMID 19282842
- [Background] Cachefo A, Boucher P, Vidon C, Dusserre E, Diraison F, Beylot M. Hepatic lipogenesis and cholesterol synthesis in hyperthyroid patients. J Clin Endocrinol Metab. 2001 Nov;86(11):5353-7. doi: 10.1210/jcem.86.11.7981. PMID 11701705
- [Background] Kassis AN, Jones PJ. Changes in cholesterol kinetics following sugar cane policosanol supplementation: a randomized control trial. Lipids Health Dis. 2008 Apr 30;7:17. doi: 10.1186/1476-511X-7-17. PMID 18447941
- [Background] Wulan SN, Westerterp KR, Plasqui G. Dietary and 24-h fat oxidation in Asians and whites who differ in body composition. Am J Clin Nutr. 2012 Jun;95(6):1335-41. doi: 10.3945/ajcn.111.031369. Epub 2012 May 2. PMID 22552026
- [Background] Adkins A, Basu R, Persson M, Dicke B, Shah P, Vella A, Schwenk WF, Rizza R. Higher insulin concentrations are required to suppress gluconeogenesis than glycogenolysis in nondiabetic humans. Diabetes. 2003 Sep;52(9):2213-20. doi: 10.2337/diabetes.52.9.2213. PMID 12941759
- [Background] Barosa C, Silva C, Fagulha A, Barros L, Caldeira MM, Carvalheiro M, Jones JG. Sources of hepatic glycogen synthesis following a milk-containing breakfast meal in healthy subjects. Metabolism. 2012 Feb;61(2):250-4. doi: 10.1016/j.metabol.2011.06.022. Epub 2011 Sep 8. PMID 21862086
- [Background] Basu A, Jensen MD, McCann F, Mukhopadhyay D, Joyner MJ, Rizza RA. Effects of pioglitazone versus glipizide on body fat distribution, body water content, and hemodynamics in type 2 diabetes. Diabetes Care. 2006 Mar;29(3):510-4. doi: 10.2337/diacare.29.03.06.dc05-2004. PMID 16505497
- [Background] Chacko SK, Sunehag AL. Gluconeogenesis continues in premature infants receiving total parenteral nutrition. Arch Dis Child Fetal Neonatal Ed. 2010 Nov;95(6):F413-8. doi: 10.1136/adc.2009.178020. Epub 2010 Aug 3. PMID 20682577
- [Background] Kao CC, Hsu JW, Bandi V, Hanania NA, Kheradmand F, Jahoor F. Resting energy expenditure and protein turnover are increased in patients with severe chronic obstructive pulmonary disease. Metabolism. 2011 Oct;60(10):1449-55. doi: 10.1016/j.metabol.2011.02.013. Epub 2011 May 6. PMID 21550084
- [Background] Letexier D, Diraison F, Beylot M. Addition of inulin to a moderately high-carbohydrate diet reduces hepatic lipogenesis and plasma triacylglycerol concentrations in humans. Am J Clin Nutr. 2003 Mar;77(3):559-64. doi: 10.1093/ajcn/77.3.559. PMID 12600843
- [Background] Money KE, Myles WS. Heavy water nystagmus and effects of alcohol. Nature. 1974 Feb 8;247(5440):404-5. doi: 10.1038/247404a0. No abstract available. PMID 4544739
- [Background] Browning JD, Burgess SC. Use of (2)H(2)O for estimating rates of gluconeogenesis: determination and correction of error due to transaldolase exchange. Am J Physiol Endocrinol Metab. 2012 Dec 1;303(11):E1304-12. doi: 10.1152/ajpendo.00306.2012. Epub 2012 Oct 2. PMID 23032685
- [Background] Vrisekoop N, den Braber I, de Boer AB, Ruiter AF, Ackermans MT, van der Crabben SN, Schrijver EH, Spierenburg G, Sauerwein HP, Hazenberg MD, de Boer RJ, Miedema F, Borghans JA, Tesselaar K. Sparse production but preferential incorporation of recently produced naive T cells in the human peripheral pool. Proc Natl Acad Sci U S A. 2008 Apr 22;105(16):6115-20. doi: 10.1073/pnas.0709713105. Epub 2008 Apr 17. PMID 18420820
- [Background] Doshi A, Zaheer A, Stiller MJ. A comparison of current acne grading systems and proposal of a novel system. Int J Dermatol. 1997 Jun;36(6):416-8. doi: 10.1046/j.1365-4362.1997.00099.x. No abstract available. PMID 9248884